CLINICAL TRIAL: NCT01891266
Title: Effects of Tourniquet Use on Physical Function and Performance in Primary Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Effects of Tourniquet Use on Physical Function and Performance in Primary Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: The Danish Rheumatism Association (Other); Bevica Fonden (Other)
Responsible Party: Principal Investigator, Rasmus Lohmann-Jensen, MSc, MSc, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-20110084
Record Dates: First submitted 2013-06-21; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-tourniquet assisted TKA (Experimental)
  Interventions: Procedure: Non-tourniquet assisted TKA
- Tourniquet assisted TKA (Other)
  Interventions: Procedure: Tourniquet assisted TKA

INTERVENTIONS:
Procedure: Non-tourniquet assisted TKA — The intervention group will undergo non-tourniquet assisted total knee arthroplasty, which means that blood flow to the lower limb is maintained throughout surgery.
  Arms: Non-tourniquet assisted TKA
Procedure: Tourniquet assisted TKA — The procedure involves the use of a tourniquet around the thigh. During surgery the tourniquet will be inflated above the systolic blood pressure to ensure a complete bloodless surgical field.
  Arms: Tourniquet assisted TKA

SUMMARY:
Background:

Osteoarthritis (OA) is the most common joint disease that causes symptomatic health problems in the elderly population. For some patients with knee OA, total knee arthroplasty (TKA) may be the only option that offers the possibility of reestablishing the patient's life quality.

Surgery of TKA usually takes place in a complete bloodless field established by a tourniquet around the thigh. The method aims to reduce blood loss and give the surgeon better visibility during the operation. The method is, however, not without side effects as patients often experience severe pain and swollen leg in the time after surgery. Furthermore, has the method shown decidedly muscle- and nerve damage followed by prolonged rehabilitation and reduced physical function.

It is, however, possible to perform the operation without the use of the tourniquet.

Aim and hypothesis:

The aim of the present study is to assess the effects of tourniquet use in TKA on physical function, early rehabilitation, pain and opioid consumption.

Hypotheses H1: TKA without tourniquet leads to better physical function and early rehabilitation.

H2: TKA without tourniquet causes less pain and opioid consumption H3: Recovery of mechanical lower limb function post TKA is faster without use of tourniquet.

Methods:

80 patients (40 in each group) all eligible for TKA will be consecutively recruited and randomized to A) TKA without tourniquet, B) TKA with tourniquet. Subjects will be evaluated before the operation (baseline) and 14 days, 3, 6 and 12 months after the operation.

The primary outcome will be the change from baseline to 3 months in self-administered knee-function (KOOS-ADL subscale). Further, will we examine a number of pre-specified secondary outcomes, which include self-rated knee-related pain, symptoms, difficulty with sports and leisure activities, and quality of life. In addition, muscle function, physical performance, and the use of pain medication will be studied

Impact of the project:

The project design of this study will enable analyses for determining the impact of operating without tourniquet and whether such an intervention can in fact improve physical function, performance and quality of life within TKA patients. The results may impact notably on the patient level and possible redefine current surgical strategies. The societal perspective of the project is to remobilize patients faster, which may reduce hospital services and absence from work.

ELIGIBILITY:
Inclusion Criteria:

* Knee Osteoarthritis both clinically and radiologically according to the "Ahlbäck classification system".
* Patients who can tolerate spinal anesthesia

Exclusion Criteria:

* Patients with rheumatoid arthritis.
* Patients with BMI > 35.
* History of major knee operations.
* Malignancy.
* Known muscle disease.
* History of deep vain thrombosis (DVT), or other blood coagulation disorders.
* Symptomatic bilateral OA, with planned surgery of the contra lateral knee within a year.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-11 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in self reported physical function. Assessed with the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire subscale for, Function in Daily Living (ADL). | Endpoint 3 months
  Further assessments: Baseline, 14 days and a 6 and 12 months follow up. KOOS is a patient-reported outcome measure with good evidence of reliability, validity and responsiveness in different population with varying pathologies, injury durations, and activity levels (http://www.koos.nu).

SECONDARY OUTCOMES:
Change in the Knee injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 14 days, 3 months (endpoint) and a 6 and 12 months follow up
  The remaining 4 subscales for pain, other symptoms, function in sport and recreation, and knee related quality of life.
Global perceived effect (GPE) score | 3 months (endpoint) and a 6 and 12 months follow up
  In addition to pain and physical function the assessment by the patient of a global perceived effect of the treatment is a recommended responder criterion [4]. Patients will be asked to rate possible change in their condition since the initial administration (baseline) on a 7-point Likert-scale.
Change in physical performance (battery). | Baseline, 3 and 14 days, 3 months (endpoint) and a 6 months follow up
  Physical performance-based measures will include; Passive knee range of motion, 30 s chair stand (number completed), 20 m normal-paced and fast-paced walk (time in sec.), and timed up and go (time in sec.)

OTHER OUTCOMES:
Change in mechanical muscle function | Baseline, 3 and 6 months
  Mechanical muscle function includes; Quadriceps strength (MVC), Rate of force development, surface electromyography, force steadiness.
Change in 30-sec Maximal Repeated Unilateral Knee Bending | Baseline, 3 and 6 months
  Measures the maximum number of knee bends performed on one leg in 30 seconds and the ability to execute fast stretch shortening cycles over the knee joint.
Change in Pain | Baseline and 1-14 days
  Self-reported pain: Pain intensity is measured using an 11-step visual analogue scale (VAS) (0 = no pain and 10 = worst possible pain). The VAS has been demonstrated to be reliable and valid in assessing the intensity of musculoskeletal knee pain [5].
  Self-reported use of pain medication: The patient's use of pain medication will be registered.
Muscle biopsies | Baseline
  Two muscle biopsy samples (2 * 100 mg) will be acquired in a subgroup of the patients (2 x 10) during operation. One sample will be collected prior to applying the tourniquet, and a second sample will be collected prior to the removal of the tourniquet. Muscle tissue is frozen in liquid nitrogen and sent for analysis at the Institute of Sports Science and Clinical Biomechanics for mechanical characteristics, Ca2+-kinetics and markers of free oxygen radicals.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Lohmann-Jensen, Cand. Scient, Principal Investigator — Odense University Hospital and University of Southern Denmark; Søren Overgaard, Professor, Study Chair — Odense University Hospital and University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Lohmann-Jensen R, Holsgaard-Larsen A, Emmeluth C, Overgaard S, Jensen C. The efficacy of tourniquet assisted total knee arthroplasty on patient-reported and performance-based physical function: a randomized controlled trial protocol. BMC Musculoskelet Disord. 2014 Mar 29;15:110. doi: 10.1186/1471-2474-15-110. PMID 24678741